CLINICAL TRIAL: NCT02340923
Title: A Device for Rapid, Painless, Bedside Muscle Evaluation of Children
Status: Completed | Type: Observational
Sponsor: Skulpt, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: PED-003-2014; 2R44NS073188 (NIH)
Record Dates: First submitted 2014-12-03; First posted 2015-01-19 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne Muscular Dystrophy; EIM
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Subjects: Healthy subjects aged 0-18 years old. Subjects cannot have a presence or past history of a neurological disorder or other disease that would be expected to substantially impact health.
- Duchenne Muscular Dystrophy Subjects: Male subjects aged 0-18 years old with genetic or histopathologic diagnosis of duchenne muscular dystrophy, or signs and symptoms of DMD and genetic or histopathologic diagnosis in a family member. Additionally, subjects cannot have the presence of a superimposed neuromuscular or other medical condition that substantially impacts the individual's health or ability to cooperate.

SUMMARY:
The purpose of this protocol is to perform Electrical Impedance Myography (EIM) testing on healthy children and children with duchenne muscular dystrophy so as to develop a new, convenient tool for the office based assessment of children with a wide variety of neuromuscular conditions.

ELIGIBILITY:
Duchenne Muscular Dystrophy:

Inclusion Criteria:

* 1. Age 0-18
* 2. Male
* 3. Genetic or histopathologic diagnosis of duchenne muscular dystrophy, or signs and symptoms of DMD and genetic or histopathologic diagnosis in a family member.

Exclusion Criteria:

* 1. Age over 18
* 2. Female
* 3. Presence of a superimposed neuromuscular or other medical condition that substantially impacts the individual's health or ability to cooperate.

Max Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Duchenne Muscular Dystrophy Subjects
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Electrical Impedance Myography Measurements | Baseline (all subjects) & 3 months, 6 months, 1 year for returning subjects only
  Up to 11 muscles will be measured using EIM technology. These muscles include: Right Lateral Deltoid, Right Biceps, Right Triceps, Right Wrist Flexors, Right Wrist Extensors, Right Vastus Lateralis, Right Tibialis Anterior, Right Gastrocnemius, Right Gluteus Medius, Right Biceps Femoris, and Right Thoracic Parapinal.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Skulpt, Inc., Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio

REFERENCES:
- [Derived] Leitner ML, Kapur K, Darras BT, Yang M, Wong B, Dalle Pazze L, Florence J, Buck M, Freedman L, Bohorquez J, Rutkove S, Zaidman C. Electrical impedance myography for reducing sample size in Duchenne muscular dystrophy trials. Ann Clin Transl Neurol. 2020 Jan;7(1):4-14. doi: 10.1002/acn3.50958. Epub 2019 Dec 25. PMID 31876124